CLINICAL TRIAL: NCT02044432
Title: Treatment of Patients With Chronic Osteoarthritis (Gonarthrosis) With Ginger Kidney Compress - a Randomized, Controlled Trial
Brief Title: Treatment of Patients With Chronic Osteoarthritis With Ginger Kidney Compress - a Randomized, Controlled Trial
Acronym: OST_02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Principal Investigator, Dr. Jan Vagedes, Dr. Jan Vagedes MD, ARCIM Institute Academic Research in Complementary and Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OST_02
Record Dates: First submitted 2014-01-10; First posted 2014-01-24 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

ARMS (2):
- Ginger compress (Experimental)
  Interventions: Other: ginger compress
- Wait list (No Intervention)

INTERVENTIONS:
Other: ginger compress — Kidney ginger compress
  Arms: Ginger compress

SUMMARY:
The investigators hypothesize that by a 5-week treatment with ginger kidney compresses at least 2 of 3 main symptoms of the WOMAC (pain, stiffness, functionality) will be reduced at least 30% at the time of the post-measurement (after 5 weeks of therapy) in comparison to the respective control group (waitlist).

ELIGIBILITY:
Inclusion Criteria:

* Chronic osteoarthritis, mainly osteoarthritis of the knee
* osteoarthritis symptoms for at least six months
* written consent to participate in the study
* Age: 30 years and more

Exclusion Criteria:

* Rheumatoid Arthritis
* Fibromyalgia
* Oncological or other serious diseases
* Use of corticosteroids
* Nephropathy
* Non-intact skin conditions in the area of application
* Hypersensitivity / allergy to ginger
* Simultaneous participation in another clinical trial

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Total Sum Score (WOMAC) | Change from baseline at 5 weeks of treatment and 5 weeks follow up

SECONDARY OUTCOMES:
Change in medication | After 5 weeks of treatment and 5 weeks follow up

OTHER OUTCOMES:
Sum Score of "Short Arthritis Assessment Scale" questionnaire | After 5 weeks of treatment and 5 weeks follow up
Parameters of a warmth questionnaire | After 5 weeks of treatment and 5 weeks follow up
Range of knee movement | After 5 weeks of treatment and 5 weeks follow up
Thermography (body heat distribution) | After 5 weeks of treatment and 5 weeks follow up